CLINICAL TRIAL: NCT03805711
Title: Transfemoral Replacement of Aortic Valve With HLT MeriDIAN Valve CE Mark Trial
Brief Title: HLT Meridian Valve CE Mark Trial
Acronym: RADIANT CE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision to stop enrollment.
Sponsor: HLT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLT 1801
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Stenosis; Transcatheter Aortic Valve Replacement; TAVR; TAVI; Aortic Valve
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Aortic Valve Replacement with HLT® Transcatheter System (Experimental): Replacement of aortic valve using the HLT® Transcatheter System (HLT System) comprised of The Meridian® II Valve with TriVent™ Anticalcification Treatment and The Pathfinder® II Delivery System
  Interventions: Device: HLT® Transcatheter System

INTERVENTIONS:
Device: HLT® Transcatheter System — Transcatheter aortic valve replacement using The HLT® Transcatheter System (HLT System) in patients with symptomatic heart disease due to severe aortic stenosis who are judged by the Heart Team to be at Intermediate or High Risk for aortic valve replacement surgery (Heart Team agrees that the risk of 30-day mortality is ≥ 3%).

SUMMARY:
To evaluate the safety and performance of the HLT System in patients with symptomatic heart disease due to severe aortic stenosis who are judged by the Heart Team to be at Intermediate or High Risk for aortic valve replacement surgery.

DETAILED DESCRIPTION:
Prospective, non-randomized, single arm, multi-center CE Mark trial.

ELIGIBILITY:
Inclusion Criteria:

* Echocardiographic or hemodynamic based evidence of severe aortic stenosis with one of the following:

  1. Aortic valve area ≤ 1.0 cm^2 or 0.6 cm^2/m^2
  2. Mean aortic valve gradient ≥ 40 mmHg
  3. Peak aortic valve velocity ≥ 4 m/sec
* Symptoms due to severe aortic stenosis resulting in one of the following:

  1. NYHA Functional Classification of II or greater
  2. Presence of angina
  3. Presence of syncope
* Documented aortic valve annular size of ≥ 24 and ≤ 26 mm (associated perimeter range is 76-81mm or associated area range of 453-530 mm2) by the MSCT Core Lab assessment of pre-procedure imaging.
* Patient is considered intermediate or high risk to undergo surgical aortic valve replacement with one of the following:

  1. Intermediate Surgical Risk: STS-PROM score of ≥ 3% to 8%
  2. High Surgical Risk: STS-PROM score of ≥ 8%
  3. Documented heart team agreement of risk for surgical aortic valve replacement (SAVR) due to other factors not captured by risk-scores (i.e. frailty or comorbidities)
* Geographically available, willing to comply with follow up and able to provide written informed consent

Exclusion Criteria:

* Patients with a coronary height of <10mm, or otherwise determined to be at high risk for coronary obstruction
* Patients with low flow/low gradient aortic stenosis
* Patients with significant annular or LVOT calcification that could compromise procedural success
* Pre-existing prosthetic heart valve in any position, or prosthetic ring
* Severe aortic, mitral or tricuspid valve regurgitation
* Untreated clinically significant coronary artery disease requiring revascularization
* Unfavorable peripheral vascular anatomy or disease (e.g. severe obstructive calcification or severe tortuosity) that would preclude passage of 18 Fr catheters from the femoral arterial access to the aorta as evidenced by peripheral MSCT
* Need for emergent surgery or intervention other than the investigational procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 days
  Freedom from all-cause mortality

SECONDARY OUTCOMES:
Procedural Device Performance | During the Procedure
  Device implant success defined as:
  Absence of procedural mortality AND, Correct positioning of a single prosthetic heart valve into the proper anatomical location AND, Intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20mmHg or peak aortic valve velocity <3 m/sec, AND no moderate or severe AR)
Post-procedural Valve Performance | 14 Days (or earlier if discharged prior to post-op Day 14), 30 Days, 6 months, 12 months, 24 months, 36 months, 48 months and 60 months
  Valve performance will be evaluated by an independent Echo Core Laboratory for the following hemodynamic parameters:
  * Aortic valve area (AVA)
  * Aortic valve regurgitation (AR)
  * Aortic valve gradient (Mean and Peak)
Rate of Adverse Events | Throughout the 5-year follow-up period, assessed annually at a minimum
  * All adverse events through the one (1) year follow up period
  * All Serious Adverse Events through the five (5) year follow up period
  * Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) at 30 Days, 6 months, 12 months and annually through five (5) years

CONTACTS AND LOCATIONS:
Overall Officials: Axel Linke, MD, Principal Investigator — Klinik für Innere Medizin und Kardiologie, Herzzentrum Dresden Universitätsklinik
Locations (1):
- Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No